CLINICAL TRIAL: NCT00183365
Title: Children of Depressed Parents: Family-Based Prevention
Brief Title: Effect of Family-Based Prevention on Children of Depressed Parents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2004-8-3934; R34MH071868 (NIH); DDTR B4-ARD
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2014-02

CONDITIONS: Depression
Keywords: Family; Parenting; Depression; Group Intervention
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Experimental): Participants will receive the Protecting Families Program with individual parent training
  Interventions: Behavioral: Parent Skills Training; Behavioral: Protecting Families Program (PFP)
- 2 (Active Comparator): Participants will receive parent training alone
  Interventions: Behavioral: Parent Skills Training

INTERVENTIONS:
Behavioral: Parent Skills Training — Parent skills training will include 10 weeks of psychoeducational and skills training group sessions for parents.
Behavioral: Protecting Families Program (PFP) — Participants will receive 10 weeks of PFP, which will include a community meal at the beginning of each session, a parent skills training group, and a concurrent cognitive behavioral therapy (CBT) group for the focal child.
  Arms: 1

SUMMARY:
This study will test the Protecting Families Program, a 10-week prevention program for depressed parents and their pre-teenage children, by comparing the effectiveness of the program versus parent training alone.

DETAILED DESCRIPTION:
Children of depressed parents are at risk for developing social-emotional problems. Despite the fact that economic hardship is a strong risk factor for both maternal depression and poor child development, little research has been conducted to develop prevention programs for low-income urban families. This randomized, open-label study will address the research gap by developing and pilot-testing the Protecting Families Program (PFP), a family-based, multi-component prevention program. The PFP will offer its services to low-income, urban, depressed parents and their children between the ages of 9 and 14.

Prior to the interventional portion of the study, several small focus groups composed of mental-health care providers and depressed parents will meet. The purpose of these focus groups will be to gather information that will help maximize the effectiveness of the remainder of the study. The interventional phase will compare PFP combined with individual parent training versus parent training alone. Participants will be randomly assigned to one of these two intervention groups. The study will last a total of 10 weeks. Both groups will meet once each week. PFP will include a community meal at the beginning of each session, a parent skills training group, and a concurrent cognitive behavioral therapy (CBT) group for the focal child. Participants' symptoms, diagnosis, functional status, family functioning, cognitive factors, and parenting practices will be assessed at the study start date, immediately post-intervention, and 6 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Parent is currently in treatment
* Parent's primary DSM-IV diagnosis is major depressive disorder, dysthymia, or depression not otherwise specified
* Parent's child lives with him/her at least part time

Exclusion criteria:

* Parent has a history or current diagnosis of any psychotic disorder or organic brain syndrome
* Parent has history of bipolar or schizoaffective disorder
* Parent's IQ is below 70
* Parent has any serious medical or neurological disorder or condition that may prevent weekly participation
* Parent has chronic pain that may prevent weekly participation
* Parent or child is currently suicidal to the extent that it will interfere with outpatient treatment
* Parent has a current substance dependence
* Child is currently seeking psychological treatment
* Child is mentally retarded (determined by school and clinic records)
* Child has a clinically severe psychiatric diagnosis

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-10; Primary Completion 2008-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Child psychiatric symptomology | Measured immediately post-treatment and at 6-month follow-up

SECONDARY OUTCOMES:
Parenting skills, family functioning, and parent social support | Measured immediately post-treatment and at 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Guy Diamond, PhD, Principal Investigator — University of Pennsylvania / CHOP; Rhonda Boyd, PhD, Principal Investigator — University of Pennsylvania / CHOP
Locations (1):
- Center for Family Intervention Science; The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States